CLINICAL TRIAL: NCT03038074
Title: Plethysmographic and Acoustic Respiration Rate Clinical Data Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BAIL0002
Record Dates: First submitted 2017-01-09; First posted 2017-01-31 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Group (Experimental): The subjects will be enrolled in the test group and will receive Pulse Oximeter with respiration rate sensor to examine the respiration rate.
  Interventions: Device: Pulse Oximeter with respiration rate sensor

INTERVENTIONS:
Device: Pulse Oximeter with respiration rate sensor

SUMMARY:
The objective of this clinical investigation is to collect high-resolution pulse oximetry, RRp, and RAM data in pediatric subjects for the purpose of algorithm optimization and to build a database of representative pulse oximetry and respiratory signal profiles for patients in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0 to 5 years old
* Fully developed skin

Exclusion Criteria:

* Subjects with skin abnormalities at the planned application sites that would interfere with sensor application.
* Subjects with pre-existing conditions and/or co-morbidities that would prohibit them from participating in the study due to unacceptable risks to their health and well-being, as determined by the Principal Investigator (PI).
* Subjects deemed not suitable for the study at the discretion of the investigator

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Collection of high-resolution pulse oximetry and RAM data in pediatric subjects | through study completion, an average of 6 months
  The objective of this clinical investigation is to collect high-resolution pulse oximetry and acoustic signals in pediatric subjects for the purpose of algorithm optimization and to build a database of representative pulse oximetry and respiratory signal profiles for patients in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Office of Mohammad T. Bailony, National City, California, United States